CLINICAL TRIAL: NCT01733511
Title: the Patients Journey Through Surgical Admission Ward Versus Emergency Department
Status: Completed | Type: Observational
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Christian Backer Mogensen, assistant professor, University of Southern Denmark
Other Study IDs: SLB-ED-03-2012
Record Dates: First submitted 2012-11-13; First posted 2012-11-27 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Waiting Time in Emergency Department

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- admitted to emergency department
- patients admitted to surgical ward

SUMMARY:
Emergency departments are established in 20 hospitals in Denmark in order to improve the quality for the acute patients.

A group of acute patients which require timely assessment and plan from a specialist is patients with abdominal pain.

the aim of the present study is to evaluate whether the admission of the group of patients to emergency departments reduces the time to doctor, specialist and plan compared to the traditional admission to a surgical acute ward.

ELIGIBILITY:
Inclusion Criteria:

* age more than 15 years

Exclusion Criteria:

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all acute admissions to hospital due to abdominal pain
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2011-02; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
time in minutes | up to 24 hours after admission
  the time in minutes from the patient is admitted until the patient is seen by a doctor and until a treatment plan is recorded

REFERENCES:
- [Derived] Schultz H, Mogensen CB, Pedersen BD, Qvist N. Front-end specialists reduce time to a treatment plan for patients with acute abdomen. Dan Med J. 2013 Sep;60(9):A4703. PMID 24001465